CLINICAL TRIAL: NCT05657496
Title: Biological Response to Platelet-rich Plasma and Corticosteroid Injections
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Principal Investigator is Retiring.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, James A. Keeney, MOI INPATIENT MEDICAL DIRECTOR, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2092036
Record Dates: First submitted 2022-07-03; First posted 2022-12-20 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Pain; Osteoarthritis; Corticosteroid; Platelet-rich Plasma (PRP)
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Triamcinolone Acetonide; Suspensions; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: The patient is randomized into one of two treatment arms. Randomization is employed using a computer-generated random assignment sequence and results kept in envelopes. The patient is blinded to the injection received. Subjects receive the injection indicated by study arm at initial visit with a synovial fluid aspiration, urine, and blood collection. At the 1-month visit, subjects provide blood, urine, and synovial fluid aspiration. After the 1-month visit if the patient is experiencing pain and wants an injection, they are instructed to schedule a visit with the PI. If an injection is indicated, the patient is unblinded to which injection they previously received and may choose which to receive. If subject received steroid injection at initial visit, they must wait 3 months before receiving another steroid injection per standard of care guidelines. Subjects is required to complete VAS, KOOS-JR, and UCLA activity surveys at baseline, 2, 4, 8, 12, 24 , 26 and 52 weeks.
Who Masked: Participant
Masking Description: Syringes will be prepared and masked with opaque tape by the clinic nurses, thus providing blinding for subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Steroid (Active Comparator): A 6mL injection at the initial visit of triamcinolone 40 mg/1 mL (Kenalog) with 5 mL of 1% lidocaine
  Interventions: Drug: Triamcinolone Acetonide 40 mg/ml Inj, Susp
- Platelet-rich Plasma (Experimental): An injection at the initial visit of approximately 4-6 mL of PRP
  Interventions: Biological: Platelet-rich plasma Inj

INTERVENTIONS:
Drug: Triamcinolone Acetonide 40 mg/ml Inj, Susp — Prepared in clinic by physician or medical staff
  Other Names: Corticosteroid injection
  Arms: Steroid
Biological: Platelet-rich plasma Inj — Produced from participant's whole blood venous draw of approximately 15 mL. Prepared by centrifuge in clinical office
  Other Names: PRP
  Arms: Platelet-rich Plasma

SUMMARY:
The goal is to determine how two different injections, corticosteroid and platelet-rich plasma, are used to treat patients with knee osteoarthritis may affect a patient's pain and function. Secondarily, the investigators are also interested in knowing how the two types of injections that will be given may affect what happens in the joint cartilage. The participants will receive one of the two injection types at the initial visit. There will be surveys to complete (around 10 questions) about the participants' knee and overall function. The investigators will ask these same questions on seven separate occasions. In addition, the investigators will ask the participants to provide blood and urine samples at our clinic before the first knee injection and before any other injection that is needed over the course of the study. During the injections, synovial fluid will be aspirated from the participants' knee at the initial visit and the one month visit. If the participants decide to go to surgery to help relieve the pain from osteoarthritis at any point during the study, the investigators will collect the material from the participants' knee that would be normally discarded as medical waste.

Previous studies have indicated that concentrations of inflammatory and degradative biomarkers in patient serum, urine, and synovial fluid may provide insight into OA pathophysiology. To our knowledge, no study has been performed to assess the impact of intra-articular PRP injection upon fluid concentrations of a comprehensive panel of proposed OA-related biomarkers. In this study, the investigators will evaluate the impact of intra-articular PRP injection upon markers of cartilage matrix turnover, inflammatory mediators, degradative enzymes, inhibitors of degradative enzymes, and markers of bone metabolism in serum, urine, and synovial fluid of knee OA patients.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is an extremely common cause of disability, with a global prevalence of 22.9% in adults aged 40 and over. OA is a whole-joint disease characterized by progressive degradation of articular cartilage, chronic inflammation of joint tissue, and subchondral bone remodeling, resulting in severe pain and decreased mobility in patients.

No cure currently exists for OA, and treatment is aimed at symptomatic management and prevention of disease progression. Currently, this consists of:

1. Initial conservative treatment for osteoarthritis across all levels of radiographic disease severity includes activity modification, oral analgesic or anti-inflammatory medications, non-supervised or supervised (e.g., physical therapy) exercise, and occasionally bracing.
2. Injection therapies have been used in the treatment of osteoarthritis for more than 60 years. Medical corticosteroids have served as a gold standard for symptom management as an intra-articular injection, but concerns have always existed around the potential for either the steroid medication (which suppresses both repair and inflammation processes) or the local anesthetic co-administered with the steroid to contribute to degradation of joint cartilage over time. Alternative substances have been developed to address the joint environment - with an intent to improve symptoms, while decreasing the potential for joint degeneration. These alternative medications include viscosupplements (hyaluronic acid analogues) and biological agents (platelet-rich plasma, or stem cell therapies).
3. Surgical interventions include arthroscopy for concurrent symptomatic meniscus tears or unstable cartilage that contribute to mechanical symptoms, osteotomy (realignment) surgery for active patients with single compartment arthritis, and arthroplasty (joint replacement) for patients with more limited activity goals, severe arthritis, and temporary-but not sustained---pain relief with the conservative treatments described in #1 and #2.

Intra-articular injection of a corticosteroid has been shown to be effective in providing short-term relief of knee OA symptoms, possibly due to anti-inflammatory and immunosuppressive effects. Repeated corticosteroid injections have thus become the standard of care for patients with mild to moderate knee OA.

Intra-articular injection of platelet-rich plasma (PRP) has emerged as a promising alternative to corticosteroid injection in knee OA patients. Studies have indicated that PRP is safe and may provide benefits such as pain relief, improved knee function, and enhanced quality of life. Moreover, PRP injection has been shown to provide longer-lasting symptomatic attenuation, with clinically significant improvement observed for as long as 12 months post-injection.

Previous studies have indicated that concentrations of inflammatory and degradative biomarkers in patient serum, urine, and synovial fluid may provide insight into OA pathophysiology. To the investigators' knowledge, no study has been performed to assess the impact of intra-articular PRP injection upon fluid concentrations of a comprehensive panel of proposed OA-related biomarkers. In this study, the investigators will evaluate the impact of intra-articular PRP injection upon markers of cartilage matrix turnover, inflammatory mediators, degradative enzymes, inhibitors of degradative enzymes, and markers of bone metabolism in serum, urine, and synovial fluid of knee OA patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 and over, presenting with a knee disorder of at least one knee
* Patients eligible for use of either corticosteroid or biological agent for treatment of moderate or severe (but not end-stage) knee osteoarthritis
* KL grade of 2-3

Exclusion Criteria:

* Subjects less than 40 years of age
* Previous reconstructive knee surgery
* Participating in another clinical trial
* Unable to receive corticosteroid injections (i.e., allergies, adverse reactions, etc.)
* Unable to sign informed consent
* Pregnant or plan to become pregnant

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Difference in concentration of MCP-1 proinflammatory biomarker from baseline in the serum after intraarticular knee injection of PRP at 1 month. | 12 months
  MCP-1 is a proinflammatory chemokine that recruits monocytes to sites of injury or inflammation. It plays a key role in the immune response and has been implicated in various chronic inflammatory and cardiovascular diseases.
Difference in concentration of MCP-1 proinflammatory biomarker from baseline in the urine after intraarticular knee injection of PRP at 1 month. | 12 months
  MCP-1 is a proinflammatory chemokine that recruits monocytes to sites of injury or inflammation. It plays a key role in the immune response and has been implicated in various chronic inflammatory and cardiovascular diseases.
Difference in concentration of MCP-1 proinflammatory biomarker from baseline in the synovial fluid after intraarticular knee injection of PRP at 1 month. | 12 months
  MCP-1 is a proinflammatory chemokine that recruits monocytes to sites of injury or inflammation. It plays a key role in the immune response and has been implicated in various chronic inflammatory and cardiovascular diseases.

SECONDARY OUTCOMES:
Difference in concentration of RANTES proinflammatory biomarker from baseline in the collected specimens after intraarticular knee injection of PRP at 1 month. | 12 months
  RANTES is a proinflammatory chemokine involved in recruiting immune cells such as T cells, eosinophils, and basophils to sites of inflammation. It plays a significant role in chronic inflammatory conditions, autoimmune diseases, and allergic responses.
Difference in concentration of IL-1b proinflammatory biomarker from baseline in the collected specimens after intraarticular knee injection of PRP at 1 month. | 12 months
  IL-1β is a key proinflammatory cytokine produced by activated macrophages and plays a central role in mediating the inflammatory response. It contributes to fever, leukocyte recruitment, and the progression of various inflammatory and autoimmune diseases.
Difference in concentration of IL-6 proinflammatory biomarker from baseline in the collected specimens after intraarticular knee injection of PRP at 1 month. | 12 months
  IL-6 is a multifunctional proinflammatory cytokine involved in immune regulation, acute phase responses, and hematopoiesis. It plays a critical role in chronic inflammation and has been associated with autoimmune disorders, infection, and cancer.
Difference in concentration of IL-8 proinflammatory biomarker from baseline in the collected specimens after intraarticular knee injection of PRP at 1 month. | 12 months
  IL-8 is a proinflammatory chemokine that primarily functions to attract and activate neutrophils at sites of infection or injury. It is involved in the pathogenesis of acute and chronic inflammatory conditions.
Difference in concentration of TNF-a proinflammatory biomarker from baseline in the collected specimens after intraarticular knee injection of PRP at 1 month. | 12 months
  TNF-α is a potent proinflammatory cytokine produced mainly by macrophages that plays a central role in systemic inflammation. It is involved in the pathophysiology of autoimmune diseases, sepsis, and chronic inflammatory conditions.
Difference in concentration of MIP-1a proinflammatory biomarker from baseline in the collected specimens after intraarticular knee injection of PRP at 1 month. | 12 months
  MIP-1α is a proinflammatory chemokine that recruits and activates immune cells, particularly monocytes, macrophages, and T cells. It plays a role in acute and chronic inflammatory responses, as well as in the progression of certain infectious and autoimmune diseases.
Difference in concentration of PGE2 proinflammatory biomarker from baseline in the collected specimens after intraarticular knee injection of PRP at 1 month. | 12 months
  PGE2 is a lipid mediator involved in the regulation of inflammation, pain, and fever through its effects on vasodilation and immune cell activity. It is produced at sites of tissue damage and contributes to both acute and chronic inflammatory responses.
Difference in concentration of IL-1RA anti-inflammatory biomarker from baseline in the collected specimens after intraarticular knee injection of PRP at 1 month. | 12 months
  IL-1RA is an anti-inflammatory cytokine that inhibits the activity of IL-1α and IL-1β by competitively binding to the IL-1 receptor without eliciting a signal. It plays a protective role in controlling excessive inflammation and is used therapeutically in inflammatory diseases like rheumatoid arthritis.
Difference in concentration of IL-4 anti-inflammatory biomarker from baseline in the collected specimens after intraarticular knee injection of PRP at 1 month. | 12 months
  IL-4 is an anti-inflammatory cytokine that promotes the differentiation of naïve T cells into Th2 cells and inhibits the production of proinflammatory cytokines. It plays a key role in regulating immune responses, particularly in allergy and humoral immunity.
Difference in concentration of IL-10 anti-inflammatory biomarker from baseline in the collected specimens after intraarticular knee injection of PRP at 1 month. | 12 months
  IL-10 is a potent anti-inflammatory cytokine that suppresses the expression of proinflammatory cytokines, chemokines, and antigen presentation. It plays a crucial role in limiting immune responses and maintaining immune homeostasis during inflammation and infection.
Difference in concentration of MMP pro-degradative biomarker from baseline in the collected specimens after intraarticular knee injection of PRP at 1 month. | 12 months
  MMPs are a family of pro-degradative enzymes that break down extracellular matrix components during normal tissue remodeling and in pathological processes. They are upregulated in inflammatory and degenerative conditions, contributing to tissue destruction and disease progression.
Difference in concentration of TIMP-1 anti-degradative biomarker from baseline in the collected specimens after intraarticular knee injection of PRP at 1 month. | 12 months
  TIMP-1 is an anti-degradative protein that inhibits matrix metalloproteinases (MMPs), helping to preserve extracellular matrix integrity. It plays a protective role in tissue remodeling and counteracts excessive degradation in inflammatory and fibrotic conditions.
Difference in concentration of TIMP-2 anti-degradative biomarker from baseline in the collected specimens after intraarticular knee injection of PRP at 1 month. | 12 months
  TIMP-2 is an anti-degradative protein that specifically inhibits several MMPs, thereby regulating extracellular matrix turnover and preventing excessive tissue breakdown. It also plays a role in modulating cell growth, angiogenesis, and tissue repair processes.
Difference in concentration of COMP from baseline in the collected specimens after intraarticular knee injection of PRP at 1 month. | 12 months
  COMP is a non-collagenous extracellular matrix protein primarily found in cartilage, tendons, and ligaments. Elevated levels in blood or synovial fluid are associated with cartilage degradation and are used as a biomarker for osteoarthritis and other joint disorders.
Difference in concentration of CTX-1 from baseline in the collected specimens after intraarticular knee injection of PRP at 1 month. | 12 months
  CTX-1 is a bone resorption marker released during the degradation of type I collagen, the main component of bone matrix. It is commonly used to assess bone turnover and monitor conditions such as osteoporosis or the effects of anti-resorptive therapies.
Difference in concentration of CTX-II from baseline in the collected specimens after intraarticular knee injection of PRP at 1 month. | 12 months
  CTX-II is a biomarker of cartilage degradation, released during the breakdown of type II collagen, which is primarily found in articular cartilage. Elevated levels are associated with joint degeneration and are commonly used in the assessment of osteoarthritis and other cartilage-related disorders.
Difference in concentration of PIICP from baseline in the collected specimens after intraarticular knee injection of PRP at 1 month. | 12 months
  PIICP is a biomarker of cartilage synthesis, released during the formation of type II collagen, a key structural component of articular cartilage. Elevated levels indicate active cartilage formation and are used to monitor cartilage repair or regeneration in joint diseases.
Difference in concentration of HA from baseline in the collected specimens after intraarticular knee injection of PRP at 1 month, and possibly 3 and 6 months timeframes | 12 months
  Hyaluronic acid is a major component of synovial fluid and extracellular matrix, playing a crucial role in joint lubrication and cartilage health. Elevated levels in serum or synovial fluid can indicate joint inflammation or degeneration, such as in osteoarthritis or rheumatoid arthritis.
Difference in concentration of biomarkers in the collected specimens after the first intraarticular knee injection of PRP from the second injection at 1 month. | 12 months
  This outcome measures the change in concentration of specific inflammatory, anti-inflammatory, degradative, and cartilage-related biomarkers in synovial fluid or blood between the first platelet-rich plasma (PRP) knee injection and the follow-up injection one month later. The goal is to assess the biological response to PRP therapy over time and identify potential markers of treatment efficacy.
Correlating the change of specific biomarker concentrations with the change of patient-reported outcome scores | 12 months
  This outcome evaluates the relationship between changes in biomarker concentrations and changes in patient-reported outcome measures (PROMs) following PRP treatment. The aim is to determine whether biological responses to therapy are associated with clinical improvements in pain, function, or quality of life.
The change From Baseline in Pain Scores on the Visual Analog Scale at 2 weeks, 4 weeks, 8 weeks, 12 weeks, 6 months, and 12 months | 12 months
  Low of 0, high of 10. Higher score means more pain and worse outcome
The change From Baseline in Scores on the UCLA Activity Score at 2 weeks, 4 weeks, 8 weeks, 12 weeks, 6 months, and 12 months | 12 months
  Low of 0, high of 10. Higher score means better knee function
The change From Baseline in Pain Scores on the Knee Injury and Osteoarthritis Outcome Score-Joint Replacement at 2 weeks, 4 weeks, 8 weeks, 12 weeks, 6 months, and 12 months | 12 months
  Multiple questions determining knee stiffness, daily functioning with knee involved activities, and knee pain.

CONTACTS AND LOCATIONS:
Overall Officials: Vicki Jones, MEd, CCRP, Study Director — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cui A, Li H, Wang D, Zhong J, Chen Y, Lu H. Global, regional prevalence, incidence and risk factors of knee osteoarthritis in population-based studies. EClinicalMedicine. 2020 Nov 26;29-30:100587. doi: 10.1016/j.eclinm.2020.100587. eCollection 2020 Dec. PMID 34505846
- [Result] Ayhan E, Kesmezacar H, Akgun I. Intraarticular injections (corticosteroid, hyaluronic acid, platelet rich plasma) for the knee osteoarthritis. World J Orthop. 2014 Jul 18;5(3):351-61. doi: 10.5312/wjo.v5.i3.351. eCollection 2014 Jul 18. PMID 25035839
- [Result] Bhatia D, Bejarano T, Novo M. Current interventions in the management of knee osteoarthritis. J Pharm Bioallied Sci. 2013 Jan;5(1):30-8. doi: 10.4103/0975-7406.106561. PMID 23559821
- [Result] Arroll B, Goodyear-Smith F. Corticosteroid injections for osteoarthritis of the knee: meta-analysis. BMJ. 2004 Apr 10;328(7444):869. doi: 10.1136/bmj.38039.573970.7C. Epub 2004 Mar 23. PMID 15039276
- [Result] Filardo G, Previtali D, Napoli F, Candrian C, Zaffagnini S, Grassi A. PRP Injections for the Treatment of Knee Osteoarthritis: A Meta-Analysis of Randomized Controlled Trials. Cartilage. 2021 Dec;13(1_suppl):364S-375S. doi: 10.1177/1947603520931170. Epub 2020 Jun 19. PMID 32551947
- [Result] Nguyen LT, Sharma AR, Chakraborty C, Saibaba B, Ahn ME, Lee SS. Review of Prospects of Biological Fluid Biomarkers in Osteoarthritis. Int J Mol Sci. 2017 Mar 12;18(3):601. doi: 10.3390/ijms18030601. PMID 28287489
- [Result] Lacko M, Harvanova D, Slovinska L, Matuska M, Balog M, Lackova A, Spakova T, Rosocha J. Effect of Intra-Articular Injection of Platelet-Rich Plasma on the Serum Levels of Osteoarthritic Biomarkers in Patients with Unilateral Knee Osteoarthritis. J Clin Med. 2021 Dec 11;10(24):5801. doi: 10.3390/jcm10245801. PMID 34945097
- [Result] Shamrock AG, Wolf BR, Ortiz SF, Duchman KR, Bollier MJ, Carender CN, Westermann RW. Preoperative Validation of the Patient-Reported Outcomes Measurement Information System in Patients With Articular Cartilage Defects of the Knee. Arthroscopy. 2020 Feb;36(2):516-520. doi: 10.1016/j.arthro.2019.08.043. Epub 2019 Dec 31. PMID 31901394
- [Result] Naal FD, Impellizzeri FM, Leunig M. Which is the best activity rating scale for patients undergoing total joint arthroplasty? Clin Orthop Relat Res. 2009 Apr;467(4):958-65. doi: 10.1007/s11999-008-0358-5. Epub 2008 Jun 28. PMID 18587624

DOCUMENTS (2):
  • Study Protocol (2022-09-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT05657496/Prot_000.pdf
  • Informed Consent Form (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT05657496/ICF_001.pdf